CLINICAL TRIAL: NCT05736965
Title: Clinical Efficacy and Safety of Selinexol Combined With Azacitidine and Venetoclax (SAV Regimen) in the Treatment of Acute Myeloid Leukemia (AML)-a Multi-center, Single-arm, Prospective Clinical Study
Brief Title: A Study of Selinexor in Combination With Azacitidine and Venetoclax (SAV Regimen) in Treatment Naïve Participants With Acute Myeloid Leukemia
Acronym: SAV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Liu Ligen, Director, Shanghai Tong Ren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAV
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: AML, Adult
Keywords: selinexor; untreated AML; azacitidine; venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAV arm (Experimental): Untreated acute myeloid leukemia who are ineligible for intensive chemotherapy or who refuse to receive intensive chemotherapy will receive selinexor in combination with azacitidine and venetoclax, 28 days per cycle, patients can receive transplants at any time once they achieved complete remission and other patients will continue to receive SAV regimen until disease progression or unacceptable toxic effects.
  Interventions: Drug: Selinexor; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Selinexor — Selinexor 60mg, PO d3,10,17
  Other Names: xpo1 inhibitor
Drug: Azacitidine — Azacitidine 75mg/m2, IV d1-3, 8-9, 15-16
Drug: Venetoclax — Venetoclax 100mg PO on day 1 and 200mg on day 2, 400mg on day 3-14
  Other Names: ABT199

SUMMARY:
This is a prospective, single-arm, multi-center clinical trial to evaluate the efficacy and safety of selinexor in combination with azacitidine and venetoclax for untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center clinical trial to evaluate the efficacy and safety of selinexor in combination with azacitidine and venetoclax for untreated acute myeloid leukemia.

Selinexor will be given orally at 60mg, d3,10,17 Azacitidine will be given at 75mg/m2, d1-3, 8-9, 15-16 Venetoclax will be given orally at 100mg on day 1 and 200mg on day 2, 400mg on day 3-14

28 days per cycle, patients can receive transplants at any time once they achieved complete remission and other patients will continue to receive treatment until disease progression or unacceptable toxic effects.

ELIGIBILITY:
Inclusion Criteria:

* Known and written informed consent voluntarily
* Age ≥ 18 years
* Newly diagnosed AML patients (per WHO 2022 classification criteria for AML diagnosis), who are not suitable for intensive chemotherapy:

  * ≥75 years or
  * Aged 18 to 74 years with at least one of the following comorbidities: Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or 3 or 4; Cardiac history of Congestive Heart Failure (CHF) requiring treatment or Ejection Fraction <= 50% or chronic stable angina; Diffusing capacity of the Lung for Carbon Monoxide (DLCO) <= 65% or Forced Expiratory Volume in 1 second (FEV1) <= 65%; Creatinine clearance >= 30 mL/min to < 45 ml/min; Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × Upper Limit of Normal (ULN); Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy .
* patients who are suitable for intensive chemotherapy but refuse it
* Liver function meets the following criteria:

aspartate aminotransferase (AST) ≤ 3.0×ULN*; alanine aminotransferase (ALT) ≤ 3.0×ULN*; Bilirubin≤1.5×ULN*; For subjects <75 years old, the bilirubin level can be ≤3.0×ULN;

* Unless due to leukemic organ involvement.

  * Renal function meets the following criteria: creatinine clearance ≥ 30 mL/min (Cockroft-Gault formula)
  * Life expectancy ≥ 4 weeks

Exclusion Criteria:

* History of any malignancies prior to study entry with exception noted in the protocol.
* Participant has known HIV infection, active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) .
* Participant has known active central nervous system (CNS) involvement with AML.
* Must not have received prior anti-AML treatment except for hydroxyurea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Composite Complete Remission | From the study start up to death (up to approximately 2 years; )
  composite complete remission(CR , CRh, CRi) was calculated based on ELN2022 criteria.

SECONDARY OUTCOMES:
overall survival (OS) | From the study start up to death (up to approximately 4 years; )
Overall response rate(ORR) | From the study start up to death (up to approximately 4 years; )
percentage of patients who achieved MRD negativity | From the study start up to death (up to approximately 4 years; )
Recurrence Free Survival(RFS) | From the study start up to death (up to approximately 4 years; )

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Changzhou Municipal No.1 People's Hospital, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - Jilin University China Japan Union Hospital, Ch’ang-ch’un
  - Harbin Institute of Hematology and Oncology, Ha’erbin
  - Anhui Provincial Hospital, Hefei
  - the first hospital of Jiaxing affiliated hospital of Jiaxing University, Jiaxing
  - Gansu Provincial People's Hospital, Lanzhou
  - Lanzhou University NO.2 Hospital, Lanzhou
  - Ningbo Medical Center Lihuili Huspital, Ningbo
  - Shanghai Ruijin Hospital, Shanghai
  - Shanghai Tong Ren hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The First Hospital of Hebei Medical University, Shijia Zhuang
  - The Second Hospital of Hebei Medical University, Shijia Zhuang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - the Second Affiliated Hospital of Wannan Medical College, Wuhu
  - Xi'an International Medical Center, Xi'an
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yixing People's Hospital, Yixing

IPD SHARING:
Plan to Share IPD: No